CLINICAL TRIAL: NCT07133178
Title: A Multicenter, Randomized, Controlled, Double-blind Pivotal Phase 3 Trial to Evaluate the Safety and Immunogenicity of a Live-attenuated Chikungunya Virus Vaccine (VLA1553) in Healthy Children Aged 1 to 11 Years
Brief Title: A Trial to Evaluate the Safety and Immunogenicity of VLA1553 in Healthy Children
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No participant recruited; trial initiation postponed to an unspecified future time while Valneva assesses potential pathways to address regulatory requests. Evaluation is ongoing to ensure alignment with regulatory expectations and obligations.
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VLA1553-322
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Chikungunya Virus Infection
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VLA1553 (Experimental): VLA1553
  Interventions: Biological: VLA1553
- Control (Active Comparator): Nimenrix will be used as Comparator
  Interventions: Biological: Control

INTERVENTIONS:
Biological: VLA1553 — Single intramuscular vaccination on Day 1 with VLA1553 full dose, a lyophilized live-attenuated Chikungunya vaccine
  Arms: VLA1553
Biological: Control — Single intramuscular vaccination on Day 1 with Nimenrix (Men ACWY vaccine), a conjugate vaccine indicated for the active immunization
  Arms: Control

SUMMARY:
VLA1553-322 is a multicenter, prospective, randomized, double-blind, phase 3 clinical trial evaluating VLA1553 in comparison to a comparator (Nimenrix®) for each stratum (age group). At least 3,000 male and female healthy children aged 1 to 11 years will be enrolled and randomized 3:1 to either VLA1553 (n=2,250) or comparator (Nimenrix®) (n=750).

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, double-blind, Phase 3 clinical trial evaluating VLA1553 in comparison to a comparator (Nimenrix®) in healthy children aged 1 to 11 years after a single vaccination in endemic countries.

The overall trial duration (First Participant In - Last Participant Out) is estimated to be approximately 22 months. Individual participation is approximately 13 months (immunogenicity subset) from ICF signature to trial completion, unless prematurely discontinued.

At least 3,000 male and female healthy children aged 1 to 11 years will be enrolled and randomized 3:1 to either VLA1553 (n=2,250) or comparator (Nimenrix®) (n=750). These children will be screened for evidence of previous CHIKV exposure.

The trial will be conducted in Latin America and / or Southeast Asia to ensure a diverse participant population and broad applicability of results. An independent Data and Safety Monitoring Board (DSMB) will oversee participant safety, review interim data, and provide recommendations on the trial's continuation. Additionally, a Valneva internal Safety Review Committee (SRC) will review safety data according to their pertinent SRC Charter.

The trial is divided into three sequential parts with predefined timepoints: Part A (Day 29, Visit 4), Part B (Month 6, Visit 6) and Part C (Month 12, Visit 7). Analyses for each part will be conducted independently after the last participant completes the respective visit, with Part A analyzed after Day 29, Part B after Month 6, and Part C after Month 12.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female healthy children aged 7 to 11 years for Stratum A, 3 to 6 years for Stratum B and 1 to 2 years for Stratum C at the time of obtaining participant informed consent / assent;
2. Written informed consent by the participant's parent(s) / Legally Acceptable Representative(s) (LAR(s), according to local requirements, and written informed assent of the participant, if applicable;
3. Participant is generally healthy as determined by the Investigator's clinical judgement based on medical history, physical examination and screening laboratory tests;
4. Participants in Stratum C (1 to 2 years) must be within the normal WHO growth and weight ranges for their age.
5. Participant is seropositive for previous CHIKV exposure (i.e. IgM+ / IgG+ or IgM- / IgG+) or seronegative (i.e. IgM- / IgG-);
6. If participant is of childbearing potential (e.g. after onset of menarche) and if involved in activities that could result in pregnancy:

   1. Female participant has a negative pregnancy test (in accordance with local regulations) at Screening (Visit 0) and Day 1 (Visit 1), respectively;
   2. Female participant has practiced an adequate method of contraception during at least the 30 days before Screening (Visit 0) and during the Screening period;
   3. Female/ male participant agrees to employ adequate birth control measures ) for the first three months post-vaccination (i.e. until Day 85, Visit 5).

Exclusion Criteria:

1. Participant who is anti-CHIKV IgM+ / IgG- does not qualify for participation in this trial.
2. Participant is taking medication or other treatment for unresolved symptoms attributed to a previous CHIKV infection; or has participated in a clinical trial involving an investigational CHIKV vaccine;
3. Participant has an acute or recent infection and who is not symptom-free in the week prior to both the Screening visit (Visit 0) and Visit 1;
4. Participant has received another live virus vaccine within 28 days or inactivated / other vaccine within 14 days prior to vaccination in this trial or plans to receive a live virus vaccine within 28 days or inactivated vaccine / other within 14 days after vaccination; Whenever possible, standard of care vaccinations should be planned with the trial VLA1553 administration in mind.
5. Participant has an ongoing medical history of or currently has acute or progressive, unstable, controlled or uncontrolled clinical condition (e.g., cardiovascular, respiratory, neurologic, psychiatric, or rheumatologic conditions) that poses a risk for participation in the trial, based on the Investigators clinical judgement. Examples include individuals with controlled, poorly controlled or unstable disease, ongoing suspected or active inflammation, or poor compliance with pharmacologic treatment, or presence of high-risk comorbidities (e.g., significant cardiopulmonary disease);
6. Participant has abnormal findings in any required trial investigations (including medical history, physical examination, and clinical laboratory) considered clinically relevant by the Investigator which pose a risk for participation in the trial based on his / her judgement;
7. Participant has a history of immune-mediated or clinically relevant arthritis / arthralgia;
8. The participant, their parent(s) / LAR(s) or siblings have a known HIV, hepatitis B or hepatitis C infection;
9. Participant has a history of malignancy;
10. Participant has a known or suspected defect of the immune system that can be expected to influence the immune response to the vaccine, such as participants with congenital or acquired immunodeficiency, including infection with HIV, status post organ transplantation or immuno-suppressive therapy within 4 weeks prior to Visit 1. Immuno-suppressive therapy is defined as administration of chronic (longer than 14 days) prednisone or equivalent ≥0.05 mg / kg / day within 4 weeks prior to trial entry, radiation therapy or immunosuppressive cytotoxic drugs / monoclonal antibodies in the previous 3 years; topical and inhaled steroids are allowed.
11. Participant has a history of any vaccine related contraindicating event (e.g., anaphylaxis, allergy to components of VLA1553 or Nimenrix®, or other known contraindications including febrile convulsions);
12. Participant presents with clinical conditions representing severe bleeding disorders and medications interfering with blood clotting;
13. Participant is pregnant (positive pregnancy test - in accordance with local regulations - at Screening or Visit 1, respectively) or is lactating at the time of enrollment or, for participants involved in activities potentially leading to pregnancy:

    1. female participants on unreliable contraception after onset of menarche
    2. male participant does not agree to employ adequate birth control measures during the first three months:
14. Participant received blood-derived products (e.g. plasma) within 180 days prior to vaccination in this trial;
15. Participant has a rash, dermatological condition or tattoos that would, in the opinion of the Investigator, interfere with injection site AE measurement and rating;
16. Participant has participated in another clinical trial involving an investigational medicinal product (IMP) or device within 30 days prior to vaccination or is scheduled to participate in another clinical trial involving an IMP, or device at any time during this trial;
17. Participant has any condition that, in the opinion of the Investigator, may compromise the participants well-being, might interfere with evaluation of trial endpoints, or would limit the participant's ability to complete the trial;
18. Participant / Participant's parent(s) / LAR(s) is / are a member of the team conducting the trial or in a dependent relationship with one of the trial team members. Dependent relationships include close relatives (i.e., children, partner / spouse, siblings, parent(s) / LAR(s) as well as employees of the Investigator or site personnel conducting the trial;
19. Participant has received the comparator (Nimenrix® or any equivalent meningococcal conjugate vaccine covering serogroups A, C, W-135, and Y) prior to the trial.

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2026-02-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants with a seroresponse as defined by μPRNT50 for baseline negative participants | 28 days post-vaccination

SECONDARY OUTCOMES:
Immune response as measured by CHIKV-specific neutralizing antibody titers as determined by μPRNT assay | on Day 1, Day 15, Day 29, Day 85, Day 180, and Month 12 (Day 365)
Proportion of participants with seroresponse as determined by μPRNT assay | on Day 15, Day 29, Day 85, Day 180 and Month 12 (Day 365)
Proportion of participants with seroconversion as compared to baseline as determined by μPRNT assay | on Day 15, Day 29, Day 85, Day 180 and Month 12 (Day 365)
Fold increase of CHIKV-specific neutralizing antibody titers determined by μPRNT assay as compared to baseline | on Day 15, Day 29, Day 85, Day 180 and Month 12 (Day 365)
Proportion of participants reaching an at least 4-fold, 8-fold, 16-fold, or 64-fold increase in CHIKV-specific neutralizing antibody titers compared to baseline as measured by μPRNT assay | on Day 15, Day 29, Day 85, Day 180 and Month 12 (Day 365)
Antibody titers, seroresponse, seroconversion and fold increases for CHIKV-specific neutralizing antibodies, determined by μPRNT assay stratified by CHIKV baseline serostatus (based on μPRNT) and age stratum | at Day 15, Day 29, Day 85, Day 180 and Month 12 (Day 365)
Frequency and severity of any Adverse Event (AE), stratified by CHIKV baseline serostatus and age stratum | until Day 29
Frequency and severity of unsolicited Adverse Events (AE), stratified by CHIKV baseline serostatus and age stratum | until Day 180 and Month 12
Frequency and severity of solicited injection site and systemic Adverse Event (AE), stratified by CHIKV baseline serostatus and age stratum | within 14 days post-vaccination
Frequency and relatedness of any Serious Adverse Event (SAE), stratified by CHIKV baseline serostatus and age stratum | during entire trial period
Frequency and severity of any adverse event of special interest (AESI), stratified by CHIKV baseline serostatus and age stratum | starting within 2 to 21 days post-vaccination
Frequency and severity of any late onset adverse event of special interest (AESI), stratified by CHIKV baseline serostatus and age stratum | during the entire trial starting 22 days post-vaccination
Frequency and severity of adverse event of special interest (AESI) (regulatory agency definition), stratified by CHIKV baseline serostatus and age stratum | with an onset within 30 days post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Valneva Clinical Development, Study Chair — Valneva Austria GmbH

IPD SHARING:
Plan to Share IPD: Yes
After trial completion, Valneva may provide access to individual de-identified participant data and related trial documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Trial Report (CTR)) upon request from qualified researchers, and subject to Valneva's review and approval.